CLINICAL TRIAL: NCT04485078
Title: The Clinical and the Functional Impact of Central Sensitization On Patients With Axial Spondyloarthritis
Brief Title: Investigation of Central Sensitization Frequency and Related Factors in Axial Spondyloarthritis Patients
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.695
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Axial Spondyloarthritis; Central Sensitisation
Keywords: Axial spondyloarthritis; central sensitization; quantitative sensory testing; central sensitization inventory
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Axial spondyloarthritis patients: QST with clinical scales
  Interventions: Diagnostic Test: Pressure pain threshold; Diagnostic Test: Temporal summation; Diagnostic Test: Conditioned pain modulation; Diagnostic Test: Central Sensitization Inventory; Other: Bath Ankylosing Spondylitis Disease Activity Index; Other: Ankylosing Spondylitis Quality of Life; Other: Istanbul Low Back Pain Disability Index; Other: Beck Depression Inventory; Other: Fatigue Severity Scale; Other: Pittsburgh Sleep Quality Index; Other: Fibromyalgia Rapid Screening Tool; Other: Visual analogue scale
- Healthy controls: QST
  Interventions: Diagnostic Test: Pressure pain threshold; Diagnostic Test: Temporal summation

INTERVENTIONS:
Diagnostic Test: Pressure pain threshold — The PPT assessments of spine will be performed over the spinous process and 2 cm right and left side of the corresponding spinous process. The regional PPT scores will be composed from sum of all PPT values for related segments at spine. The sacroiliac PPT scores will be obtained bilaterally from four measurement points; the first point is located 1 cm medially and caudally from spina iliaca posterior superior (SIPS) and 3 more laterally, medially and cranially.The left trapezius muscle will be used to evaluate distant control point .The 1 cm2 algometer probe will be placed vertically in the each selected point and pressure will be increased with 0.1 kg/sc until the participant reporting pressure became painful. The pressure value at which the pain is first felt will be accepted as the PPT of that point.
  Other Names: PPT
Diagnostic Test: Temporal summation — TS will be evaluated over the trapezius muscle, sacroiliac joints, C7, T6, and L3 levels at spine with manuel algometer. TS scores will be calculated for each spine level as the sum of three values which measured over the spinous process and 2 cm right and left side of corresponding level. In the evaluation of TS, a pressure as much the PPT value of each point will be applied with pain pressure algometer ten times with a 1-second interstimulus interval. Patients will be asked to rate their pain using on a 0 to 10 visual analogue scale (VAS) at 0, 5, and 10 seconds. TS will be calculated by subtracting the rating at 0 seconds from the rating at 10 seconds. The point that is located 1 cm medially and caudally from SIPS was used for SI joint TS measurement on both sides.
  Other Names: TS
Diagnostic Test: Conditioned pain modulation — First stimulus will be applied to trapezius with the pressure that induced a pain intensity of 4 point on a 10 point VAS as called a test stimulus. After that the right hand of the patient will be immersed in 70C water for 20 seconds to create a conditioning stimulus. Second test stimulus with the same intensity of first one will be applied to trapezius after the conditioning stimulus and patients will be asked to rate their pain. If the patients cannot hold their hand in the water for 20 seconds, the test stimulus will be applied immediately after the patients removed their hands out of water. The ratio between the first and second VAS values multiplied by 100 will be defined as CPM score
  Other Names: CPM
  Groups: Axial spondyloarthritis patients
Diagnostic Test: Central Sensitization Inventory — Standardized questionnaire to determine the level of central sensitization
  Other Names: CSI
  Groups: Axial spondyloarthritis patients
Other: Bath Ankylosing Spondylitis Disease Activity Index — Standardized questionnaire to determine the level of disease activity in AxSpa patients
  Other Names: BASDAI
  Groups: Axial spondyloarthritis patients
Other: Ankylosing Spondylitis Quality of Life — Standardized questionnaire to investigate the quality of life in AxSpa patients
  Other Names: ASQoL
  Groups: Axial spondyloarthritis patients
Other: Istanbul Low Back Pain Disability Index — Standardized questionnaire to investigate the disability
  Other Names: ILPBDI
  Groups: Axial spondyloarthritis patients
Other: Beck Depression Inventory — Standardized questionnaire to investigate the depression
  Other Names: BDI
  Groups: Axial spondyloarthritis patients
Other: Fatigue Severity Scale — Standardized questionnaire to investigate the fatigue
  Other Names: FSS
  Groups: Axial spondyloarthritis patients
Other: Pittsburgh Sleep Quality Index — Standardized questionnaire to investigate the sleep quality and disturbance
  Other Names: PSQI
  Groups: Axial spondyloarthritis patients
Other: Fibromyalgia Rapid Screening Tool — Standardized questionnaire to detect fibromyalgia
  Other Names: FIRST
  Groups: Axial spondyloarthritis patients
Other: Visual analogue scale — global pain score on a 0 to 10
  Other Names: VAS
  Groups: Axial spondyloarthritis patients

SUMMARY:
The term axial spondyloarthritis (axSpA) describes a group of chronic inflammatory diseases that characterized with spinal involvement. AxSpA is one of the most common rheumatic diseases and chronic pain and morning stiffness are the main complaints of these patients. Central sensitization is defined as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with many rheumatological diseases has been demonstrated in several studies. Pain in axSpA patients is generally considered as a result of increased inflammatory burden and structural changes, However, failure to adequate analgesia in every patient whose inflammation is suppressed with anti-inflammatory treatment suggests new pain mechanisms. Central sensitization (CS) is one of these mechanisms and its recognition is only possible by detailed evaluation of the patient. There is no method for the diagnosis of central sensitization is accepted as a gold standard. clinical scales and quantitative sensory testing (QST) widely is used for this purpose widely. The most commonly used QST types include pressure pain threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM). The well-known scale used for the evaluation of central sensitization is the Central Sensitization Inventory , developed by Mayer et.al in 2011 for detect central sensitization in chronic pain patients. The aim of this study is to evaluate the frequency of central sensitization (CS) in patients with axSpA by means of clinical scales and quantitative sensory testing (QST), to examine related comorbidities and the parameters associated with the development of sensitization in these patients.

DETAILED DESCRIPTION:
The term axial spondyloarthritis (axSpA) describes a group of chronic inflammatory diseases that characterized with spinal involvement. AxSpA is one of the most common rheumatic diseases and chronic pain and morning stiffness are the main complaints of these patients. Central sensitization (CS) is defined as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with many rheumatological diseases has been demonstrated in several studies. However, data associated with central sensitization in axSpA patients is very limited. The quantitative sensory testing (QST) is commonly used for detection hyperalgesia and allodynia those are accepted main findings in sensitized patients. The most commonly used QST types include pressure pain threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM).Pressure pain threshold measurement is frequently used to show local / generalized sensitivity increase in patients who develop pain sensitization. For this purpose, the pain response of superficial or deep tissue can be evaluated through mechanical device called algometer. The algometer probe was placed vertically in the each selected point and pressure was increased until the participant reporting pressure became painful. The first pressure value at which pain is felt is considered the PPT of that point. TS is defined as a progressive increase in pain response with repetitive painful stimuli. This condition is also known as wind-up phenomenon and play a role to development CS. CPM, known as one of the main mechanisms of endogenous analgesia, is based on the principle that pain perception can be reduced with painful stimulus applied to different areas according to the "pain inhibits pain" model. In the CPM testing, it is aimed to investigate the modulator effect of two different painful stimuli on each other. The diagnosis of CS can be made with QST or with Central Sensitization Inventory (CSI). The aim of this study is to evaluate the frequency of central sensitization (CS) in patients with axial spondyloarthritis (AxSpA) by means of clinical scales and quantitative sensory testing (QST), to examine related comorbidities and the parameters associated with the development of sensitization in these patients. The patients with AxSpa and healthy controls will be included in this study. QST which consists of pressure pain threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM) will be applied to the patient and control groups. Disease activity (BASDAI), functional status (ASQoL, ILBPDI), sleep quality (PSQI), pain (VAS pain), depression (BDI) and fatigue (FSS) will be assessed. Fibromyalgia (FIRST) and other comorbidities will be investigated. Patients will be divided as the ones with and without CS according to the central sensitization inventory (CSI) and the results will be compared. After data collection, analysis will be performed with the appropriate statistical method

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with axSpA according to the Assessment of SpondyloArthritis International Society (ASAS) criteria Aged between 18-65 years

Exclusion Criteria:

Had an other rheumatic diseases, peripheral vascular disease, peripheral neuropathy and spine disease (e.g., symptomatic herniated disc, spinal stenosis), Using centrally acting pain medications (e.g., pregabaline, duloxetine, opioids) or glucocorticoids (>10 mg prednisone or its equivalent) within 3 months of study enrollment

The exclusion criteria of the control grup were same as that of the patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients aged 18-65 years diagnosed with axSpA according to the ASAS criteria will be recruited from a Rheumatology outpatient clinic of a single tertiary care hospital
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | 3 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points.

SECONDARY OUTCOMES:
Pressure pain threshold | 3 months
  The spinal hyperalgesia will be evaluated from C3 and C7 (cervical); T6 and T2 (thoracic); L3 and L5 (lumbar) levels. The PPT assessments of these levels were performed over the spinous process and 2 cm right and left side of the corresponding spinous process. The sacroiliac PPT scores were obtained from four measurement points [1]. Trapezius muscle will be used to evaluate distant control point
Temporal summation | 3 months
  TS scores will be evaluated over the trapezius muscle, sacroiliac joints, C7, T6, and L3 spine. TS scores will be calculated for each spine as the sum of three values which measured over the spinous process and 2 cm right and left side of corresponding level. In the evaluation of TS, a pressure as much the PPT value of each point will be applied with pain pressure algometer ten times with a 1-second interstimulus interval. Patients will ve asked to rate their pain using visual analogue scale (VAS) at 0, 5, and 10 seconds. TS will be calculated by subtracting the rating at 0 seconds from the rating at 10 seconds
Conditioned pain modulation | 3 months
  For the assessment of conditioned pain modulation (CPM), first stimulus will be applied to trapezius with the pressure that induced a pain intensity of 4 point on a 10 point VAS. After that the right hand of the patient will be immersed in 7 degrees Celcius water for 20 seconds to create a conditioning stimulus. Second stimulus with the same intensity of first one was applied to trapezius after the conditioning stimulus and patients asked to rate their pain. The ratio between the first and second VAS values will be defined as CPM
VAS pain | 3 months
  The patients pain severity will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 3 months
  BASDAI is one of the most frequently used scales for determining disease activity in axSpA patients and includes questions to evaluate the patient's axial and peripheral symptoms, fatigue and morning stiffness. The questionnaire consists of 10 questions in total and is interpreted in favor of disease activity of 4 points or more.
Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) | 3 months
  This scale was developed by Doward et.al in 2003 and consists of 18 questions in total. Each question is answered as yes or no, and the total score is calculated by evaluating the yes answer as 1 and no as 0. It is frequently used in clinical practice because it helps to evaluate the effects of the disease and determine treatment strategies in patients diagnosed with AxSpa.
Istanbul Low Back Pain Disability Index (ILBPDI) | 3 months
  This scale was developed for assessing the severity of disability in chronic low back pain patients by Duruöz et.al in 2013. This scale consists of 18 questions in the form of a Likert scale that evaluates the limitation of daily life activities of patients in the last month.
Beck Depression Inventory (BDI) | 3 months
  This questionnaire consists of 21 questions, each with four options. Scoring is interpreted as 0-9 normal, 10-18 mild depression, 19-29 moderate depression and 30-63 points as severe depression.
Fatigue severity scale (FSS) | 3 months
  The FSS includes 9 questions included in order to determine the negative effects of fatigue intensity and fatigue on daily life activities in the last week. İf the score more than 6.1, this is interpreted in favor of chronic fatigue syndrome.
Pittsburgh Sleep Quality Index (PSQI) | 3 months
  This scale is designed for quantitative measurement of sleep quality and consists of 24 questions in total. The questions are divided into 7 sections those included sleep disturbance-related symptoms. High scores are associated with poor sleep quality.
Fibromyalgia Rapid Screening Tool | 3 months
  This questionnaire is consisted of 6 questions in which fibromyalgia-related clinical parameters are investigated. The patient scoring at least 5 points is considered has fibromyalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet T DURUOZ, Professor, Study Chair — Marmara University
Locations (1):
- Feyza Nur YUCEL, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Strand V, Singh JA. Patient Burden of Axial Spondyloarthritis. J Clin Rheumatol. 2017 Oct;23(7):383-391. doi: 10.1097/RHU.0000000000000589. PMID 28937474
- [Result] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Result] Arendt-Nielsen L, Graven-Nielsen T, Svensson P, Jensen TS. Temporal summation in muscles and referred pain areas: an experimental human study. Muscle Nerve. 1997 Oct;20(10):1311-3. doi: 10.1002/(sici)1097-4598(199710)20:103.0.co;2-5. PMID 9324089
- [Result] Yarnitsky D, Bouhassira D, Drewes AM, Fillingim RB, Granot M, Hansson P, Landau R, Marchand S, Matre D, Nilsen KB, Stubhaug A, Treede RD, Wilder-Smith OH. Recommendations on practice of conditioned pain modulation (CPM) testing. Eur J Pain. 2015 Jul;19(6):805-6. doi: 10.1002/ejp.605. Epub 2014 Oct 20. PMID 25330039
- [Result] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Result] Doward LC, Spoorenberg A, Cook SA, Whalley D, Helliwell PS, Kay LJ, McKenna SP, Tennant A, van der Heijde D, Chamberlain MA. Development of the ASQoL: a quality of life instrument specific to ankylosing spondylitis. Ann Rheum Dis. 2003 Jan;62(1):20-6. doi: 10.1136/ard.62.1.20. PMID 12480664
- [Result] Duruoz MT, Ozcan E, Ketenci A, Karan A. Development and validation of a functional disability index for chronic low back pain. J Back Musculoskelet Rehabil. 2013;26(1):45-54. doi: 10.3233/BMR-2012-00349. PMID 23411648
- [Result] van Leeuwen RJ, Szadek K, de Vet H, Zuurmond W, Perez R. Pain Pressure Threshold in the Region of the Sacroiliac Joint in Patients Diagnosed with Sacroiliac Joint Pain. Pain Physician. 2016 Mar;19(3):147-54. PMID 27008288
- [Result] Middlebrook N, Heneghan NR, Evans DW, Rushton A, Falla D. Reliability of temporal summation, thermal and pressure pain thresholds in a healthy cohort and musculoskeletal trauma population. PLoS One. 2020 May 29;15(5):e0233521. doi: 10.1371/journal.pone.0233521. eCollection 2020. PMID 32469913
- See also: IASP terminology — https://www.iasp-pain.org/Education/Content.aspx?ItemNumber=1698#Centralsensitization